CLINICAL TRIAL: NCT01317576
Title: Optimizing the Beneficial Health Effects of Exercise for Diabetes: Focus on the Liver!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bram Brouwers (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Bram Brouwers, Drs, Maastricht University Medical Center
Organization: Maastricht University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 11-3-002
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity
Keywords: Magnetic Resonance Spectroscopy; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity; Motor Activity

ARMS (3):
- Healthy control (Experimental): This group will exist of healthy obese that are matched for BMI and age with the type 2 diabetes group and non-alcoholic fatty liver disease group.
  Interventions: Behavioral: Exercise intervention
- Non-alcoholic fatty liver disease (Experimental): This group will exist of people that suffer from non-alcoholic fatty liver disease. They will be matched for BMI and age according to the Type 2 diabetes group
  Interventions: Behavioral: Exercise intervention
- Type 2 diabetes patients (Experimental): This group will exist of patients that suffer from type 2 diabetes
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — Subjects will be training for 12 week, 3 times a week. Two times a week they will perform a 30 minutes bicycle training. Once a week they will perform a 30 minutes resistance training.

SUMMARY:
Due to the western lifestyle, correlated with a high calorie intake and low physical activity, obesity is becoming a major health problem. All over the world obesity reaches epidemic proportions. Obesity is closely linked to type 2 diabetes, a multi-factorial disease that increases the presence of multiple health problems. Until now, exercise and dietary intervention seem to be the single most effective interventions to treat obesity and type 2 diabetes mellitus. In obesity and type 2 diabetes, not only fat accumulation in adipose tissue, but also fat accumulation in the peripheral tissues occurs. Fat accumulation in peripheral tissues has been associated with insulin resistance. Exercise seems to have a positive effect on the accumulation of fat in the peripheral tissue and on the insulin sensitivity in type 2 diabetic patients.

In this study we want to investigate if a prolonged exercise training program can lower the intrahepatic lipid content and can improve the metabolism of the liver in type 2 diabetic patients and patients with non-alcoholic fatty liver disease, and to examine if this leads to improvements in metabolic risk markers. To this end, we will include investigation of the effect of exercise on adipose tissue (inflammatory markers and adipocyte size) and skeletal muscle (ex vivo lipid metabolism) to incorporate the effect of exercise on liver, muscle and adipose tissue and to clarify the crosstalk between these tissues in the pathophysiology of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects:

   * Male sex
   * Age 40-70 years
   * BMI 27-35 kg/m2
   * Stable dietary habits
   * Sedentary: No participation in any kind of sports for at least 2 years.
2. For diabetic patients only:

   * Must be on sulphonylurea or metformin therapy for at least 6 months with constant dose for at least 2 months, or on a dietary treatment for at least 6 months
   * Well-controlled diabetes: fasting plasma glucose concentration ≥ 7.0 mmol/l and < 10.0 mmol/l at the time of screening.
3. For subjects with non-alcoholic fatty liver disease:

   * Liver fat content ≥ 5,56%, based on the formula of Kotronen et al. and confirmed with MRS.
   * Fasting plasma glucose concentration must be < 7.0 mmol/l
4. For control subjects:

   * Liver fat content < 5,56%, based on the formula of Kotronen et al. and confirmed with MRS.
   * Normoglycemic according to the WHO criteria (OGTT)

Exclusion Criteria:

1. All subjects:

   * Female sex
   * Unstable body weight (weight gain or loss > 3 kg in the past three months)
   * Participation in an intensive weight-loss program or in vigorous exercise program during the last year before the start of the study.
   * Active cardiovascular disease. (This will be determined by questionnaires and by screening on medication. Furthermore, all subjects will undergo a physical examination by a medical doctor).
   * Chronic renal dysfunction (creatinine > 2 increased (normal values: 64-104 µmol/l))
   * Use of Thiazolidines (glitazone/rosiglitazone/pioglitazone/troglitazone)
   * Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg
   * Haemoglobin < 7.5 mmol/l (anaemia)
   * Blood donor
   * Use of medication known to interfere with glucose homeostasis (i.e. corticosteroids), except for diabetic patients.
   * Use of anti-thrombotic medication
   * Claustrophobia and contra-indications for MRI
   * Abuse of alcohol(> 3 units (1unit = 10 gram ethanol) per day)
   * Abuse of drugs
   * Participation in another biomedical study within 1 month before the first screening visit
2. For diabetics:

   * Severe diabetes which requires application of insulin or patients with diabetes-related complications
3. For controls:

   * Liver disease or liver dysfunction (ALAT > 2.5 x increased)

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proton Magnetic resonance spectroscopy to measure the reduction in liver fat content after a training intervention | 16 weeks
Magnetic resonance spectroscopy to measure the ATP and Pi concentrations in the liver | 16 weeks
13C-methionine breath test to measure hepatic mitochondrial function | 16 weeks
  Subjects will drink a solution of 200ml H2O with 13C-Methionine. The following 2 hours, every 10 minutes a breath sample will be taken and analysed to measure the concentration of 13C in the exhaled breath.
Euglycemic-hyperinsulinemic clamp for measurement of insulin sensitivity and metabolic flexibility | 16 weeks
  After taking fasting blood samples, a primed constant infusion of glucose is initiated. Plasma glucose levels are clamped at ~5 mmol/L by variable co-infusion of 20 % glucose. Every 5 minutes, blood is sampled for immediate determination of plasma glucose concentration. Glucose infusion rate is adjusted to obtain plasma glucose levels of ~5 mmol/L (euglycemia). A bolus of insulin is then infused. Before and during steady state, substrate oxidation is measured using an indirect calorimeter, which determines metabolic flexibility.
Blood sampling to determine the concentration of cardiovascular risk factors in the blood before and after exercise | 16 weeks

SECONDARY OUTCOMES:
Peripheral arterial tonometry to measure endothelial function, as a marker for cardiovascular risk. | 16 weeks
Echography of the heart to measure diastolic dysfunction | 16 weeks
Fat biopsy to measure adipose tissue inflammatory markers and adipocyte size before and after training intervention | 16 weeks
  A small amount of abdominal subcutaneous adipose tissue (~1g) will be collected under local anaesthesia (2% lidocain) using needle biopsy (with the needle connected to a vacuum syringe). Inflammatory markers in the adipose tissue (e.g. IL-6, IL-8, IL-1b, PAI-1, TNFa, CD68, CD163, CD11b, MCP-1, leptin, adiponectin mRNA expression) and adipocyte size will be analysed
Muscle biopsy to measure muscle mitochondrial density, muscle mitochondrial function and muscle lipid metabolism | 16 weeks
  . After local anaesthesia (2.0% Xylocain without adrenaline), a 5-mm diameter side-cutting needle will be passed through a 7-mm skin incision, according to the protocol of the Medical Ethical committee of the Academic Hospital and University of Maastricht. The muscle biopsy will be used to measure ex vivo lipid metabolism, muscle mitochondrial density and muscle mitochondrial function.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Study Director — Maastricht University; Bram MW Brouwers, M.S., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Kotronen A, Peltonen M, Hakkarainen A, Sevastianova K, Bergholm R, Johansson LM, Lundbom N, Rissanen A, Ridderstrale M, Groop L, Orho-Melander M, Yki-Jarvinen H. Prediction of non-alcoholic fatty liver disease and liver fat using metabolic and genetic factors. Gastroenterology. 2009 Sep;137(3):865-72. doi: 10.1053/j.gastro.2009.06.005. Epub 2009 Jun 12. PMID 19524579
- [Background] Meex RC, Schrauwen-Hinderling VB, Moonen-Kornips E, Schaart G, Mensink M, Phielix E, van de Weijer T, Sels JP, Schrauwen P, Hesselink MK. Restoration of muscle mitochondrial function and metabolic flexibility in type 2 diabetes by exercise training is paralleled by increased myocellular fat storage and improved insulin sensitivity. Diabetes. 2010 Mar;59(3):572-9. doi: 10.2337/db09-1322. Epub 2009 Dec 22. PMID 20028948
- [Background] Kelley DE, McKolanis TM, Hegazi RA, Kuller LH, Kalhan SC. Fatty liver in type 2 diabetes mellitus: relation to regional adiposity, fatty acids, and insulin resistance. Am J Physiol Endocrinol Metab. 2003 Oct;285(4):E906-16. doi: 10.1152/ajpendo.00117.2003. PMID 12959938
- [Derived] Vanweert F, Boone SC, Brouwers B, Mook-Kanamori DO, de Mutsert R, Rosendaal FR, Lamb HJ, Schrauwen-Hinderling VB, Schrauwen P, Hesselink MKC, Phielix E. The effect of physical activity level and exercise training on the association between plasma branched-chain amino acids and intrahepatic lipid content in participants with obesity. Int J Obes (Lond). 2021 Jul;45(7):1510-1520. doi: 10.1038/s41366-021-00815-4. Epub 2021 May 2. PMID 33935282
- [Derived] Mancilla R, Brouwers B, Schrauwen-Hinderling VB, Hesselink MKC, Hoeks J, Schrauwen P. Exercise training elicits superior metabolic effects when performed in the afternoon compared to morning in metabolically compromised humans. Physiol Rep. 2021 Jan;8(24):e14669. doi: 10.14814/phy2.14669. PMID 33356015
- [Derived] Stinkens R, Brouwers B, Jocken JW, Blaak EE, Teunissen-Beekman KF, Hesselink MK, van Baak MA, Schrauwen P, Goossens GH. Exercise training-induced effects on the abdominal subcutaneous adipose tissue phenotype in humans with obesity. J Appl Physiol (1985). 2018 Nov 1;125(5):1585-1593. doi: 10.1152/japplphysiol.00496.2018. Epub 2018 Sep 13. PMID 30212302
- [Derived] Brouwers B, Schrauwen-Hinderling VB, Jelenik T, Gemmink A, Havekes B, Bruls Y, Dahlmans D, Roden M, Hesselink MKC, Schrauwen P. Metabolic disturbances of non-alcoholic fatty liver resemble the alterations typical for type 2 diabetes. Clin Sci (Lond). 2017 Jul 7;131(15):1905-1917. doi: 10.1042/CS20170261. Print 2017 Aug 1. PMID 28620012